CLINICAL TRIAL: NCT03527069
Title: Phase III, National, Multicenter, Randomized, Double Blind Clinical Trial, to Evaluate the Efficacy and Safety of Cipros 10 Association on Dyslipidemia Treatment
Brief Title: Efficacy and Safety of Cipros 10 Association on the Isolated Hypertriglyceridemia and Dyslipidemia Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0617-CIPROS
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Hypertriglyceridemia; Dyslipidemia
MeSH Terms: conditions — Hypertriglyceridemia; Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIPROS 10 (Experimental): The study is double-Masked, the patient wil take 2 tablets, as follow:
  1 tablet Cipros 10 association; and
  1 tablet crestor placebo Oral, once a day.
  Interventions: Drug: Cipros 10 association
- Crestor (Active Comparator): The study is double-Masked, the patient wil take 2 tablets, as follow:
  1 tablet Crestor 10mg; and
  1 tablet Cipros association placebo Oral, once a day.
  Interventions: Drug: Crestor 10 mg

INTERVENTIONS:
Drug: Cipros 10 association — oral, once a day.
  Other Names: EMS association
  Arms: CIPROS 10
Drug: Crestor 10 mg — oral, once a day.
  Other Names: Rosuvastatin 10 mg
  Arms: Crestor

SUMMARY:
The purpose of this study is to evaluate the efficacy of Cipros 10 association in the treatment of Dyslipidemia Treatment

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes, aged 18 years or more;
* Participants with the diagnosis of Dyslipidemia presentinf low or intermediate cardiovascular risk, according to the Brazilian Guidelines on Dyslipidemia and Prevention of Atherosclerosis;
* Signed consent.

Exclusion Criteria:

* Diagnosis of familial hypercholesterolemia and other genetic diseases;
* Using medications that may interfere with the metabolism or serum levels of triglycerides;
* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* Presence of concomitant cardiovascular disease, renal failure and hepatic Failure;
* Decompensated diabetes;
* Current smoking;
* History hypersensitivity to the active ingredients used in the study;
* Pregnancy or risk of pregnancy and lactating patients;
* History of alcohol abuse or illicit drug use;
* Participation in clinical trial in the year prior to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Reduction of serum triglyceride levels measured between the first visit and last visit. | 12 weeks

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study. | 13 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Allergisa, Campinas, São Paulo, Brazil